CLINICAL TRIAL: NCT02515734
Title: A Randomized Phase II Study to Investigate the Deepness of Response of FOLFOXIRI Plus Cetuximab (Erbitux) Versus FOLFOXIRI Plus Bevacizumab as the First-line Therapy in Metastatic Colorectal Cancer Patients With RAS Wild-type Tumors: DEEPER
Brief Title: A Study of FOLFOXIRI Plus Cetuximab vs. FOLFOXIRI Plus Bevacizumab
Acronym: DEEPER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Japan Clinical Cancer Research Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JACCRO CC-13
Record Dates: First submitted 2015-07-12; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer
Keywords: FOLFOXIRI; Bmab; Cmab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOXIRI+Bmab (Active Comparator): Patients in the FOLFOXIRI + Bmab group receive until 12 cycles of FOLFOXIRI plus bevacizumab, consisting of a 30-minute infusion of bevacizumab at a dose of 5 mg per kilogram, a 60-minute infusion of irinotecan at a dose of 150 mg per square meter, and a 120-minute infusion of oxaliplatin at a dose of 85 mg per square meter and a concomitant 120-minute infusion of leucovorin at a dose of 200 mg per square meter, followed by a 48-hour continuous infusion of fluorouracil to a total dose of 2400 mg per square meter. Cycles were repeated every 14 days. After 13 cycles, patients receive fluorouracil, leucovorin and bevacizumab every 14 days until disease progression.
  Interventions: Drug: fluorouracil; Drug: Leucovorin; Drug: irinotecan; Drug: oxaliplatin; Biological: bevacizumab
- FOLFOXIRI+Cmab (Experimental): Patients in the experimental group received until 12 cycles of FOLFOXIRI plus cetuximab, consisting of a 30-minute infusion of cetuximab first time at a dose of 400 mg per kilogram, after the second time at a dose of 250mg per kilogram, a 60-minute infusion of irinotecan at a dose of 150 mg per square meter, and a 120-minute infusion of oxaliplatin at a dose of 85 mg per square meter and a concomitant 120-minute infusion of leucovorin at a dose of 200 mg per square meter, followed by a 48-hour continuous infusion of fluorouracil to a total dose of 2400 mg per square meter. Cycles were repeated every 14 days. After 13 cycles, patients receive fluorouracil, leucovorin and cetuximab every 14 days until disease progression.
  Interventions: Drug: fluorouracil; Drug: Leucovorin; Drug: irinotecan; Drug: oxaliplatin; Biological: cetuximab

INTERVENTIONS:
Drug: fluorouracil
  Other Names: 5-fluorouracil; 5-FU
Drug: Leucovorin
  Other Names: Levofolinate
Drug: irinotecan
  Other Names: CPT-11
Drug: oxaliplatin
  Other Names: eloxatin
Biological: bevacizumab
  Arms: FOLFOXIRI+Bmab
Biological: cetuximab
  Arms: FOLFOXIRI+Cmab

SUMMARY:
This study is to verify the advantage of FOLFOXIRI plus cetuximab over FOLFOXIRI plus bevacizumab as the first-line therapy in metastatic colorectal cancer patients with RAS wild-type tumors.

DETAILED DESCRIPTION:
This study is to verify the advantage of FOLFOXIRI plus cetuximab over FOLFOXIRI plus bevacizumab as the first-line therapy in metastatic colorectal cancer patients with RAS wild-type tumors. In this study the investigators employed deepness of response as a primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer
* RAS wild-type
* Measurable lesion by RECIST (Ver.1.1)
* No past history of chemotherapy in the case of unresectable primary lesion/distant metastasis/lymph node metastasis.In the case of recurrence, no treatment for the first recurrence lesion after operation
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-1.The case >=71 years is PS0.
* Life expectancy of more than 6 months
* Patients have enough organ function for study treatment within 14 days before enrollment;

  1. White blood cell (WBC)>=3,000/mm3, <12,000/mm3.
  2. Neu>=1,500/mm3.
  3. Platelet count (PLT) >=10.0x104/mm3.
  4. Hb>=9.0g/dL.
  5. Total Bilirubin<=1.5x Upper Limited Normal (ULN)
  6. aspartate aminotransferase (AST) <=2.5xULN.
  7. alanine aminotransferase (ALT) <=2.5xULN.
  8. Creatinine<=1.5xULN.
  9. Proteinuria<=1+.
  10. prothrombin time-international normalized ratio (PT-INR) <=1.5
* Must be able to swallow tablets
* Written informed consent

Exclusion Criteria:

* Synchronous multiple malignancy or metachronous multiple malignancy within 5 years disease free interval
* Lynch syndrome
* Brain metastases
* Infectious disease
* Interstitial lung disease or pulmonary fibrosis
* Comorbidity or history of serious heart failure
* History of thromboembolic events
* Cerebrovascular disease
* History of hemoptysis/hematemesis
* Uncontrolled hypertension (systolic BP>180mmHg, or diastolic BP>100mmHg)
* Sensory alteration or paresthesia interfering with function
* Large quantity of pleural, abdominal or cardiac effusion
* Severe comorbidity (renal failure, liver failure, hypertension, etc)
* Prior radiotherapy for primary and metastases leision
* Men/women who are unwilling to avoid pregnancy
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test
* History of severe allergy
* HBsAg positive or active viral hepatitis
* Administration of blood products/ Granulocyte-Colony Stimulating Factor (G-CSF), and blood transfusion within 14 days
* Surgical procedure or such as skin-open biopsy, trauma surgery, or other more intensive surgery within 28 days
* Systematic administration of antiplatelet drug or non steroid anti-inflammatory drugs (NSAIDs)
* Diathesis of bleeding (history of hemoptysis, including cavitation and/or necrosis in lung metastasis confirmed by imaging), coagulopathy
* History of gastrointestinal perforation within 1 year
* Unhealed traumatic bone fracture
* Uncontrolled diarrhea
* History of organ recipient
* Prior cetuximab/bevacizumab/Irinotecan/Oxaliplatin treatment (Adjuvant therapy by Oxaliplatin is excluded)
* Administration of atazanavir sulfate
* Jaundice
* Ileus or bowel obstruction
* Clinical diagnosis of Alzheimer's Disease
* Insulin dependent diabetes
* Thyroid disease
* Any other cases who are regarded as inadequate for study enrollment by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Best deepness of response | up to 2 years
  The maximum tumor shrinkage rates by Response Evaluation Criteria in Solid Tumors (RECIST) throughout the treatments

SECONDARY OUTCOMES:
Early tumor shrinkage | at 8 weeks
  The rates of tumor shrinkage by RECIST at 8 weeks
Response rate | up to 2 years
Deepness of response | at 4 months
  The tumor shrinkage rates by RECIST at 4 months
Overall survival | up to 2 years
Progression free survival | up to 2 years
Rate of curatively resected metastatic lesion | up to 2 years
Number of adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Toshifusa Nakajima, MD, Study Director — Japan Clinical Cancer Research Organization